CLINICAL TRIAL: NCT02841462
Title: Hydrothermal Ablation in Recurrent and Chronic Symptomatic Bursitis With the Ablaflex Device: An Open, Exploratory, 6-month Dose-tolerance and Dose Response Study
Brief Title: Hydrothermal Ablation in Recurrent and Chronic Symptomatic Bursitis
Acronym: VMT-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vesalius Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMT-001
Record Dates: First submitted 2016-06-10; First posted 2016-07-22 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Bursitis
Keywords: thermal ablation; recurrent Bursitis; chronic Bursitis; olecranon; intra-bursal perfusion
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bursitis (Experimental): Intra-bursal thermal ablation
  Interventions: Device: Intra-bursal thermal ablation

INTERVENTIONS:
Device: Intra-bursal thermal ablation — A single 3-minute intra-bursal perfusion of a physiological saline solution at increasing temperatures using the Ablaflex device.
  Other Names: Ablaflex

SUMMARY:
The overall objective of this trial is to explore the dose-tolerance (safety) and dose-response (efficacy) of single 3-minute intra-bursal perfusions of a physiological saline solution at increasing temperatures.

DETAILED DESCRIPTION:
This is an open, exploratory, 6-months dose-tolerance and dose-response study of a single thermal ablation (Ablaflex) procedure in subjects suffering from chronic symptomatic bursitis.

Possible study participants will be screened for eligibility based on defined inclusion and exclusion criteria.

Eligible patients will be administered with a single 3-minute perfusion of a physiological saline solution at a specific temperature between 50° Celsius and 55° Celsius. If the volume of the bursa estimated by ultrasound examination is ≤ 10 cc, the perfusion will be performed at a rate of 3mL/second. If the volume of the bursa is > 10 cc and ≤ 25 cc, the perfusion will be performed at a rate of 4mL/second. If the volume of the bursa is > 25 cc, the subject is considered as screen failure (exclusion criterion # 10). Immediately prior to and immediately after the thermal ablation phase of 3 minutes, perfusion with a physiological saline solution at room temperature (22°C) will be performed during 2 minutes. In total the bursa will be rinsed during 7 minutes. An elastic bandage (Elastoplast) will be applied immediately after the procedure to compress the bursa cavity. It should be worn for 6 weeks.

The first patient with bursitis of olecranon will be administered physiological saline solution at a temperature of 50° Celsius, and subsequent patients will receive perfusions with increments of 0.5 to 1° Celsius as long as no AR (of any intensity) is reported.

As long as no AR is reported, but when a first CR or PR is reported for a specific temperature, the patient in whom CR or PR was reported will be considered as the first in a cohort of 3 patients treated at the same temperature during the course of the clinical trial.

As soon as a first AR is reported, the patient in whom the AR was reported will be considered as the first in a cohort of 3 patients treated at the same temperature and the remainder of the study will be conducted with cohorts of 3 patients treated in the same conditions.

Patients will be assessed at 6 different study visits: at baseline (Day 1), 1 day (24/72h) after treatment, 1 week after treatment (+/- 1 day), 3 weeks after treatment (+/- 2 days), 6 weeks (+/- 1 week) after treatment, and 6 months (+/- 2 weeks) after treatment. At any time during the 6-months study period an unscheduled visit may be performed. Patients will be requested to score weekly patient reported outcome assessments (PRO) until Week 6 and at Month 6, and to record any possible ARs and bursitis related treatments. At Week 2, Week 4 and Week 5 the patient will complete the PRO at home.

Assessments to be performed at every study visit include: physical examination (with focus on the bursitis), vital signs (including HR and temperature), PRO, adverse events (AE), concomitant medication(s) and treatment(s). An ultrasound exam of the bursa (according to standard ultrasound protocol) is to be performed at baseline and at week 6 (week 1 assessment is optional).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
2. Subject is fluent in Dutch and is able to read and understand study documents, such as the informed consent form, patient reported outcomes and diaries.
3. Subject understands the investigational nature of the trial and is willing and able to comply with the trial requirements.
4. Subject is aged ≥ 18 years.
5. Subject is suffering from a recurrent bursitis of the olecranon, trochanter, prepatellar or infrapatellar region, confirmed by ultrasound examination (with image), or from a chronic (>6 weeks) first episode bursitis of these regions.

Exclusion Criteria:

1. Subject is pregnant or nursing.
2. Subject has fever (>37.5°C), a septic bursitis (confirmed by suppurative aspirate or positive bacteriagram), or an infection or inflammation (other than bursitis related) of the associated joint.
3. Subject has previously received corticoid drug treatment for his/her bursitis within 1 month from baseline.
4. Subject suffers from non-bursitis related pain that may, according to the investigator, interfere with bursitis-related pain assessment.
5. Subject may not, according to the investigator, be able to participate or comply reliably with study procedure requirements (due to e.g. any psychiatric disorder).
6. Subject suffers from a dermatological or other disease that may interfere with the study, its procedures and the study treatment administration (use of needles) or anesthetic procedures.
7. Subject suffers from insulin dependent diabetes or a clinically relevant blood clotting disorder.
8. Subject receives immunotherapy, chemotherapy, immunodepressant treatment, or systemic corticosteroid treatment (locally administered corticosteroids, except in the bursitis region, and inhaled corticoid treatments are allowed).
9. Subject is planning to move or travel in the next 6 months, which will interfere with or jeopardize the study follow-up schedule.
10. Bursa volume estimated by ultrasound examination > 25 cc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05-01; Primary Completion 2022-12 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Bursitis related disability as assessed on Patient Reported Outcome (PRO) | From Baseline to week 6
  Patient Reported Outcome (PRO) form assesses change from baseline on week 6. The PRO form will consist of the DASH (DASH: Disabilities of the Arm, Shoulder and Hand) for olecranon bursitis.

SECONDARY OUTCOMES:
Bursa volume as assessed with ultrasound examination | From Baseline to Week 6
  Ultrasound examination assesses response to treatment by measuring change of bursa volume at week 6 compared to baseline, resulting in either Complete Response (CR), Partial Response (PR), Minor Response (MR) No Response (NR) as defined in the protocol
Bursa volume as assessed with ultrasound examination | From Baseline to Month 6
  Ultrasound examination assesses response to treatment by measuring change of bursa volume at month 6 compared to baseline, resulting in either Complete Response (CR), Partial Response (PR), Minor Response (MR) No Response (NR) as defined in the protocol
Patient treatment satisfaction as assessed with Patient Global Impression (PGI) | From Baseline to Week 6
  Patient Global Impression (PGI) form assesses change from baseline at 6 weeks after treatment
Patient treatment satisfaction as assessed with Patient Global Impression (PGI) | From Baseline to Month 6
  Patient Global Impression (PGI) form assesses change from baseline at 6 months after treatment
Physician treatment satisfaction as assessed with Clinical Global Impression (CGI) Efficacy Index | Week 1
  Clinical Global Impression (CGI) Efficacy Index assesses, for each treatment, the perceived safety and efficacy of the study treatment administered (investigator) after treatment
Physician treatment satisfaction as assessed with Clinical Global Impression (CGI) Efficacy Index | Week 3
  Clinical Global Impression (CGI) Efficacy Index assesses, for each treatment, the perceived safety and efficacy of the study treatment administered (investigator) after treatment
Physician treatment satisfaction as assessed with Clinical Global Impression (CGI) Efficacy Index | Week 6
  Clinical Global Impression (CGI) Efficacy Index assesses, for each treatment, the perceived safety and efficacy of the study treatment administered (investigator) after treatment
Physician treatment satisfaction as assessed with Clinical Global Impression (CGI) Efficacy Index | Month 6
  Clinical Global Impression (CGI) Efficacy Index assesses, for each treatment, the perceived safety and efficacy of the study treatment administered (investigator) after treatment
Bursitis related disability as assessed on Patient Reported Outcome (PRO) | From Baseline to day 1
  Patient Reported Outcome (PRO) form assesses change from baseline on day 1. The PRO form will consist of the DASH (DASH: Disabilities of the Arm, Shoulder and Hand) for olecranon bursitis.
Bursitis related disability as assessed on Patient Reported Outcome (PRO) | From Baseline to Week 2
  Patient Reported Outcome (PRO) form assesses change from baseline on week 2. The PRO form will consist of the DASH (DASH: Disabilities of the Arm, Shoulder and Hand) for olecranon bursitis.
Bursitis related disability as assessed on Patient Reported Outcome (PRO) | From Baseline to Week 3
  Patient Reported Outcome (PRO) form assesses change from baseline on Week 3. The PRO form will consist of the DASH (DASH: Disabilities of the Arm, Shoulder and Hand) for olecranon bursitis.
Bursitis related disability as assessed on Patient Reported Outcome (PRO) | From Baseline to Month 6
  Patient Reported Outcome (PRO) form assesses change from baseline on month 6. The PRO form will consist of the DASH (DASH: Disabilities of the Arm, Shoulder and Hand) for olecranon bursitis.

OTHER OUTCOMES:
Bursa examination as assessed with Anamnesis and Physical examination | week 1
  A complete physical examination will be performed on each participant.
Bursa examination as assessed with Anamnesis and Physical examination | week 3
  A complete physical examination will be performed on each participant.
Bursa examination as assessed with Anamnesis and Physical examination | week 6
  A complete physical examination will be performed on each participant.
Bursa examination as assessed with Anamnesis and Physical examination | 6 months
  A complete physical examination will be performed on each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Berghs, MD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- Vesalius Medical Technologies, Hoegaarden, Belgium

IPD SHARING:
Plan to Share IPD: No